## The University of New Mexico Health Sciences Center **Consent to Participate in Research**

## Clinical Action of Curcumin/Turmeric in Chronic Subdural Hematoma Recurrence (CACTIS)

8/29/2018

#### Introduction

This consent form is written to address a research subject. If you will be providing permission as a legally authorized representative, the words 'you' and 'your' should be read as 'the research subject.'

You are being asked to participate in a research study being done by Dr. Howard Yonas and his associates in the Department of Neurosurgery, who propose to study a common food spice, **curcumin**, as a treatment for patients with subdural hematomas.

Subdural hematoma (SDH) is a collection of blood between two layers of tissue surrounding but not in the brain. Bleeding occurs between the dura, the outer layer and the arachnoid, the inner layer. The blood is under the skull and but not in the brain itself. As blood accumulates, however, pressure in the brain increases, which can cause neurologic symptoms that can be life-threatening.

SDH commonly occur after traumatic brain injury (TBI). It is a challenging neurosurgical problem because it often requires repeated surgical removal, with additional complications and costs for the patient and the hospital.

Surgery and removal of the blood is effective but no method for preventing the recurrence of the bleed in chronic subdural hematoma (cSDH) is available. We hope to develop a treatment to prevent the recurrence of the cSDH after surgery by treatment, with curcumin.

Studies showed that markedly increased levels of IL-8, an injury chemical in the brain, occurs in the hematoma fluid, which could be responsible for bleeding. The common cooking spice, curcumin is a potent **inhibitor** of IL-8, and it may be effective in preventing recurrence of cSDH after surgical removal of the blood. Curcumin, derived from the dietary spice turmeric, shows a wide range of beneficial effects, one being as an anti-inflammatory medication. Studies in animals and humans have shown that curcumin is extremely safe even at very high doses.

You are being asked to participate in this study because you have been clinically diagnosed with a unilateral cSDH (head bleed on one side of your head).

48 patients, of which you will be one, with unilateral cSDH, who have consented for surgery for removal of the blood, will be recruited. 24 will be treated orally with a plabeco pill, and 24 will be treated with Curcumin.

This form will explain the research study and the possible risks and benefits to you. We encourage you to talk with your family and friends before you decide to take part in this research study. If you have any questions, please ask one of the study investigators.

### What will happen if I decide to participate?

If you agree to take part in this study, you will have to do the following:

- Go to all scheduled visits, which is the standard of care visit.
- Follow the study staff's instructions about the study
- Tell the study staff about all of your medical history. This is for your own safety.
- Tell the study staff about any side effects, illnesses, problems or injuries that occur
- Tell the study staff if you plan to have any surgery or any other medical treatment or procedure.
- During the study, you may not be allowed to take certain medications. This includes prescription, over-the-counter and/or herbal medications.
- You should talk to the study staff before taking any new medication during the study.

You will be randomly assigned to one of two study groups either 1) the placebo arm or 2) the curcumin arm. You will begin by taking the pill within 48 hours after surgery. You will take one capsule three times a day for 60 days. You will undergo standard post-operative care with regard to surgery, imaging and clinical follow-up as described below. All procedures, including CT scans, are routine standard of care (SOC) in our clinic.

### **CT Imaging:**

- Post-operative day one CT scan (SOC)
- Post subdural drain removal CT scan (SOC)
- If the subdural has not resolved, you will receive an additional CT scan (SOC) for an appointment one month following the previous appointment (Approximately postoperative day 37)
  - o This will continue on a monthly basis for 6 months until resolution of blood clot.
  - o Resolution will be defined as total residual subdural cavity volume of 80cc or less.
- If the clot resolves, you don't have to come back for follow up visits, and you will be asked to give back the rest of your pills.
- During the surgery to evacuate the blood: we will remove 10 cc of the fluid that is obtained from the cSDH clot to study the inflammatory factors (IL-8) and other molecules, along with 5 cc of blood from an existing intravenous line to be used in laboratory studies.
  - o Chronic subdural fluid removed during initial surgery (10 cc of fluid/per patient), and 5 cc blood simultaneously from an existing IV.

### How long will I be in this study?

Participation in this study will be 6 months.

What are the risks or side effects of being in this study?

Except for the addition of the study drug/placebo, the management and follow-ups are all standard of care (SOC) for all cSDH patients seen by the UNM Neurosurgery department. The risks of surgery and radiation exposure from CT scans of the head are already well documented and are SOC.

The study drug curcumin (CC) is an active ingredient in the popular cooking spice turmeric. CC used for this study is concentrated into a single capsule. Known possible adverse effects of the supplement include headache, skin rash, upset stomach, abdominal pain, nausea, and diarrhea, which were seen to resolve within 1-3 days, but no other adverse effects were identified up to doses of 8 grams. There are no known adverse risks or known drug interactions with curcumin and black pepper but there may be unforeseeable risks that remain unknown.

There are risks of stress, emotional distress, inconvenience and possible loss of privacy and confidentiality associated with participating in a research study.

For more information about risks and side effects, ask the investigator.

### What are the benefits to being in this study?

There is no known benefit to the participation in this study, however, the purpose of this study is to investigate whether curcumin reduces the recurrence of surgically drained cSDH and prevent the growth of already existing subdural hematomas.

Curcumin has been extensively studied for other possible medical benefits including the reduction of cholesterol, pain from osteoarthritis, and management of other inflammatory diseases.

### What other choices do I have if I do not want to be in this study?

Your participation in this study is voluntary. You can decide not to be in the study and you can change your mind about being in the study at any time. There will be no penalty to you, and you won't lose any benefits except for benefits having to do with the study. Your regular medical care at University of New Mexico Hospital will not change if you decide not to be in the study. If you want to stop being in the study, tell the study doctor or study staff.

The study doctor can remove you from the study at any time, even if you want to stay in the study. This could happen if:

The study doctor believes it is best for you to stop being in the study.

You do not follow directions about the study.

If you stop being in the study early, the study doctor or study staff may ask you some questions about being in the study. To help you leave the study safely, the study doctor may ask you to participate in more tests.

#### How will my information be kept confidential?

We will take all possible measures to protect the security of all your personal information, but there is a small risk of loss of privacy.

Information will be entered into your study file and into a secure computer database without using your name or other information which would specifically identify you. A study number will be assigned, and a link between your name and your study number will be kept (for the purpose of follow up) in a secure drive on the researcher's computer. Medical information created by this study may be a part of your medical record.

Information contained in your study records is used by study staff and, in some cases it will be shared with the sponsor of the study. The University of New Mexico Health Sciences Center Human Research Review Committee (HRRC) that oversees human subject research, and the Food and Drug Administration and/or other entities may be permitted to access your records. There may be times when we are required by law to share your information. However, your name will not be used in any published reports about this study. A copy of this consent form will also be kept in your medical record and another copy will be provided to you.

### What are the costs of taking part in this study?

While you are in the study, you still need to get regular medical care. You (and/or your health care payer) will still have to pay for the costs of your regular medical care that are not a part of this study. You **do not** have to pay for study drug (curcumin or placebo).

## What will happen if I am injured or become sick because I took part in this study?

If you are injured or become sick as a result of this study, UNMHSC will provide you with emergency treatment, at your cost.

No commitment is made by the University of New Mexico Health Sciences Center (UNMHSC) to provide free medical care or money for injuries to participants in this study.

In the event that you have an injury or illness that is caused by your participation in this study, reimbursement for all related costs of care will be sought from your insurer, managed care plan, or other benefits program. If you do not have insurance, you may be responsible for these costs. You will also be responsible for any associated co-payments or deductibles required by your insurance.

It is important for you to tell the investigator immediately if you have been injured or become sick because of taking part in this study. If you have any questions about these issues, or believe that you have been treated carelessly in the study, please contact the Human Research Review Committee (HRRC) at the University of New Mexico Health Sciences Center, Albuquerque, New Mexico 87131, (505) 272-1129 for more information.

## Will I be paid for taking part in this study?

You will not be paid for taking part of the study.

### How will I know if you learn something new that may change my mind about participating?

You will be informed of any significant new findings that become available during the course of the study, such as changes in the risks or benefits resulting from participating in the research or new alternatives to participation that might change your mind about participating.

CACTIS Trial 5

### Can I stop being in the study once I begin?

Your participation in this study is completely voluntary. You have the right to choose not to participate or to withdraw your participation at any point in this study without affecting your future health care or other services to which you are entitled.

The study doctor can remove you from the study at any time, even if you want to stay in the study. This could happen if:

The study doctor believes it is best for you to stop being in the study.

You do not follow directions about the study.

## HIPAA Authorization for Use and Disclosure of Your Protected Health Information (HIPAA)

As part of this study, we will be collecting health information about you and sharing it with others This information is "protected" because it is identifiable or "linked" to you.

#### **Protected Health Information (PHI)**

By signing this Consent Document, you are allowing the investigators and other authorized personnel to use your protected health information for the purposes of this study. This information may include: results of physical exams, medical history, etc.

In addition to researchers and staff at UNMHSC and other groups listed in this form, there is a chance that your health information may be shared (re-disclosed) outside of the research study and no longer be protected by federal privacy laws. Examples of this include disclosures for law enforcement, judicial proceeding, health oversight activities and public health measures.

#### **Right to Withdraw Your Authorization**

Your authorization for the use and disclosure of your health information for this study shall not expire unless you cancel this authorization. Your health information will be used or disclosed as long as it is needed for this study. However, you may withdraw your authorization at any time provided you notify the UNM investigators in writing. To do this, please send letter notifying them of your withdrawal to:

Dr. Howard Yonas MSC 10 5615 1 University of New Mexico Albuquerque New Mexico 87131

Please be aware that the research team will not be required to destroy or retrieve any of your health information that has already been used or shared before your withdrawal is received.

#### Refusal to Sign

If you choose not to sign this consent form and authorization for the use and disclosure of your PHI, you will not be allowed to take part in the research study

### Subjects who are unable to consent and their Legal Authorized Representative (LAR) **Initially consented:**

In case subject will not be able to consent for the study, then the investigator and clinical team will assess these patients for capacity and identify the LAR. If the individual regains capacity during participation, the study will be explained to her/him, and she/he can decide whether continue participation.

#### Where can I find Information about this study?

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. The link is:

## https://clinicaltrials.gov/ct2/show/NCT02469857?term=AB103&rank=1

#### Whom can I call with questions or complaints about this study?

If you have any questions, concerns or complaints at any time about the research study, Dr. Howard Yonas, or his associates will be glad to answer them at 505-272-6094.

If you need to contact someone after business hours or on weekends, please call patient advocate at 505-272-0943

If you would like to speak with someone other than the research team, you may call the UNMHSC HRRC at (505) 272-1129.

## Whom can I call with questions about my rights as a research participant?

If you have questions regarding your rights as a research participant, you may call the UNMHSC HRRC at (505) 272-1129. The HRRC is a group of people from UNM and the community who provide independent oversight of safety and ethical issues related to research involving human participants. For more information, you may also access the HRRC website at http://hsc.unm.edu/som/research/hrrc/.

CACTIS Trial 7

# **CONSENT**

| You are making a decision whether to participate in this study. Your signature below indicates that |
|---|
| you read the information provided (or the information was read to you). By signing this consent |
| form, you are not waiving any of your legal rights as a research participant. |

| 11 7 1 | ons and all questions have been answered to participate in this study. A copy of thi | 2 |
|---|---|---|
| Name of Adult Subject (print) | Signature of Adult Subject | Date |
| Legally Authorized Representative (print) | Signature of Legally Authorized Representative | Date |
| | rticipant and answered all of his/her ques<br>described in this consent form and | |
| Name of Investigator/ Research Team | Member (type or print) | |
| (Signature of Investigator/ Research T | Feam Member) Date | |